CLINICAL TRIAL: NCT04808193
Title: European Perioperative Brugada Survey
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EUPerBrugadaSurvey
Record Dates: First submitted 2021-02-12; First posted 2021-03-22 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-03

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brugada Survey (Experimental): Survey will be answered by all participants
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Participants will fill in the survey

SUMMARY:
The aim of this survey is to assess the current perception and clinical practice of Resident and Board-certified Anaesthesiologists and Intensivists regarding perioperative care of patients burdened with the Brugada Syndrome. It is intended to investigate this primarily on national and secondarily on European level.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have received an invitation to participate in the survey through the online platform of the European Society of Anaesthesiology and Intensive Care.

Exclusion Criteria:

* Uninvited participation in the survey is not possible.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire about treatments for Brugada patients | 1 hour
  Number of participants with treatment-related information as assessed by the survey/questionnaire N/A

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided